CLINICAL TRIAL: NCT01684943
Title: Selecting Insulin Analogs for Closed-Loop Control Using Multiplex Pharmacokinetic Profiling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010P001005
Record Dates: First submitted 2012-08-21; First posted 2012-09-13 (Estimated); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes
Keywords: Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: All subjects participated in the single arm of the study. Some subjects participated in the continuous insulin monitoring sub-study in addition to the main protocol, or separate from the main protocol.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiplex pharmacokinetic profiling (Experimental): Multiplex pharmacokinetic profiling of regular human insulin, insulin aspart, insulin lispro, insulin glulisine, and regular human insulin. All subjects participated in the single study arm and received injections of each type of insulin. Blood samples were drawn at intervals for pharmacokinetic profiling.
  Interventions: Other: Multiplex pharmacokinetic profiling
- Continuous insulin monitoring (Experimental): Continuous insulin monitoring (CIM) of insulin lispro. Some subjects participated in the CIM sub-study, which is distinct from the Multiplex Pharmacokinetic Profiling study. This intervention involved administering insulin lispro and monitoring pharmacokinetic profile of the drug using blood samples and an investigational continuous insulin monitoring system.
  Interventions: Other: Continuous insulin monitoring

INTERVENTIONS:
Other: Multiplex pharmacokinetic profiling
  Arms: Multiplex pharmacokinetic profiling
Other: Continuous insulin monitoring
  Arms: Continuous insulin monitoring

SUMMARY:
The investigators are doing this research study to compare the pharmacokinetics (PK) (rate of absorption) of insulin lispro (Humalog), insulin aspart (Novolog), and insulin glulisine (Apidra) within individual subjects.

Additionally, the investigators will perform a preliminary feasibility evaluation of a minimally invasive continuous insulin monitoring (CIM) device and its use to derive PK parameters in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older with clinical type 1 diabetes for at least five years
* Diabetes managed using an insulin infusion pump and rapid- or very-rapid-acting insulins including insulin aspart (NovoLog), insulin lispro (Humalog), and insulin glulisine (Apidra).
* Ability to consume a sufficient amount of carbohydrates over 2-3 hours to cover 9 units of rapid acting insulin

Exclusion Criteria:

* Unable to provide informed consent
* Unable to comply with study procedures
* Inadequate venous access as determined by study nurse or physician at time of screening.
* Pregnancy
* History of gastric banding, gastric bypass, or other gastrointestinal condition that may prevent a subject from consuming a normal sized meal
* Hemoglobin <13.5 for men, < 12 for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-07; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 enrolled in Multiplex PK profiling, 9 were ineligible. 21 completed.
  3 enrolled in the CIM arm of the trial. 2 completed, 1 was excluded from analysis.
  1 subject enrolled in both study phases. They completed the MultiPK profiling experiments, but were excluded from the CIM analysis.
  Total protocol enrollment was 33.
Groups:
- Multiplex Pharmacokinetic (PK) Profiling: Multiplex pharmacokinetic profiling of regular human insulin, insulin aspart, insulin lispro, insulin glulisine, and regular human insulin
  Multiplex pharmacokinetic profiling
- Continuous Insulin Monitoring (CIM): Continuous insulin monitoring of insulin lispro
  Continuous insulin monitoring
- Multiplex PK Profiling and Continuous Insulin Monitoring: Subjects that participated in both the multiplex PK profiling experiments and the continuous insulin monitoring experiments
Period: Overall Study
Arm/Group | Multiplex Pharmacokinetic (PK) Profiling | Continuous Insulin Monitoring (CIM) | Multiplex PK Profiling and Continuous Insulin Monitoring
Started | 29 | 3 | 1
Completed | 20 | 2 | 0
Not Completed | 9 | 1 | 1
Not completed — Inadequate Venous Access | 3 | 0 | 0
Not completed — Principal Investigator Determination | 1 | 0 | 0
Not completed — Excluded from Analysis | 1 | 1 | 1
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Planning Pregnancy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Multiplex Pharmacokinetic Profiling: Multiplex pharmacokinetic profiling of regular human insulin, insulin aspart, insulin lispro, insulin glulisine, and regular human insulin
  Multiplex pharmacokinetic profiling
- Continuous Insulin Monitoring: Continuous insulin monitoring of insulin lispro
  Continuous insulin monitoring
- Multiplex PK Profiling and Continuous Insulin Monitoring: Participated in both study phases, the multiplex PK profiling visits and the CIM visits
- Total: Total of all reporting groups
Arm/Group | Multiplex Pharmacokinetic Profiling | Continuous Insulin Monitoring | Multiplex PK Profiling and Continuous Insulin Monitoring | Total
Number analyzed (Participants) | 29 | 3 | 1 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.09 (14.83) | 37.97 (26.40) | 74.65 | 47.09 (16.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 1 | 19
  Male | 14 | 0 | 0 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 25 | 2 | 1 | 28
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 26 | 2 | 1 | 29
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 3 | 1 | 25

OUTCOME MEASURES:

1. Primary Outcome: For Multiplex PK Profiling: Aggregate Mean Difference in Tmax Between the Analog With Greatest and the Analog With the Least Value of Tmax for Individuals
Description: The average difference in tmax between lispro and aspart in all participants
Time Frame: 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes after dose
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- All Participants: All participants who completed the MultiPK visits
Arm/Group | All Participants
Number analyzed (Participants) | 21
minutes | 24.28 (41.29)

2. Primary Outcome: For Continuous Insulin Monitoring: Time to Maximum Plasma Insulin and Time to Maximum Continuous Insulin Monitoring Insulin
Time Frame: 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes after dose
Population: Only 2 of the 4 experiments conducted under the Continuous Insulin Monitoring sub-study protocol produced usable data for analysis. Those two experiments are both reported here
Measure: Number; unit: minutes
Groups:
- Experiment #3: This includes the data from experiment #3. Only 2 of the 4 experiments conducted under the Continuous Insulin Monitoring sub-study protocol produced usable data for analysis. Those two experiments are both reported here.
- Experiment #4: This includes the data from experiment #4. Only 2 of the 4 experiments conducted under the Continuous Insulin Monitoring sub-study protocol produced usable data for analysis. Those two experiments are both reported here.
Arm/Group | Experiment #3 | Experiment #4
Number analyzed (Participants) | 1 | 1
minutes
  Plasma insulin tmax | 40 | 60
  CIM insulin tmax | 44 | 106

3. Secondary Outcome: Multiplex PK: Average Baseline HbA1c Categorized According to Baseline Use of Insulin Analog Found to Have the Most Favorable PK Profile for Each Individual
Description: Subjects with a difference in tmax between analogs will be categorized as follows: using insulin with best PK for them, using insulin with worst PK for them, or using insulin with intermediate PK for them. The average A1c for each of the three categories is reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Participants Using the Faster Insulin: Participants who were using the insulin analog at baseline that we determined had a faster tmax for this individual
- Participants Using the Slower Insulin: Participants who were using the insulin analog at baseline that we determined had a slower tmax for this individual
- Participants Where the Two Insulins Were the Same: Participants who we determined had no difference in the tmax between the two analogs
Arm/Group | Participants Using the Faster Insulin | Participants Using the Slower Insulin | Participants Where the Two Insulins Were the Same
Number analyzed (Participants) | 5 | 2 | 14
percentage of glycosylated hemoglobin | 8.1 (1.1) | 8.6 (1.8) | 7.5 (1.1)

4. Secondary Outcome: Multiplex PK: Count of Subjects With Difference in Tmax Between the Analog With Greatest and the Analog With the Least Value of Tmax That is > 25%
Time Frame: 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 140, 160, 180, 200, 220, 240, 260, 280, 300 minutes after dose
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 21
Participants | 11

5. Secondary Outcome: Multiplex PK: Average Baseline HbA1c Categorized According to Baseline Use of Insulin Analog With Tmax < 60 Minutes vs. Use of an Insulin Analog With Tmax > 60 Minutes for Each Individual
Description: Subjects with a difference in tmax between analogs will be categorized as follows: using insulin with tmax less than or equal to 60 minutes or using insulin with tmax > 60 minutes. The average A1c per group is reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Subjects Using Insulin With a Tmax < 60 Minutes: Participants who were using the insulin analog at baseline that we determined had a tmax of less than 60 minutes for this individual.
- Subjects Using Insulin With a Tmax of > 60 Minutes: Participants who were using the insulin analog at baseline that we determined had a tmax of more than 60 minutes for this individual.
Arm/Group | Subjects Using Insulin With a Tmax < 60 Minutes | Subjects Using Insulin With a Tmax of > 60 Minutes
Number analyzed (Participants) | 20 | 1
percentage of glycosylated hemoglobin | 7.8 (1.2) | 7.3 (NA) — Only one subject used an insulin analog at baseline that had a tmax > 60 minutes, so no standard deviation calculation is possible

6. Secondary Outcome: Multiplex PK: Average Number of Hypoglycemia Events Over the Last Month at Baseline Categorized According to Baseline Use of Insulin Analog Found to Have the Most Favorable PK Profile for Each Individual
Description: Subjects with a difference in tmax between analogs will be categorized as follows: using insulin with best PK for them, using insulin with worst PK for them, or using insulin with intermediate PK for them. The average number of hypoglycemic events per month per group is reported.
Time Frame: 1 month prior to study entry
Measure: Mean (Standard Deviation); unit: events in the month prior to study entry
Arm/Group | Participants Using the Faster Insulin | Participants Using the Slower Insulin | Participants Where the Two Insulins Were the Same
Number analyzed (Participants) | 5 | 2 | 14
events in the month prior to study entry | 8.6 (12.1) | 15.0 (15.6) | 13.1 (13.9)

ADVERSE EVENTS:
Time Frame: During the 5-hour in-clinic visits, visits occurred over the course of 1 year on average
Groups:
- Multiplex Pharmacokinetic Profiling Only: Multiplex pharmacokinetic profiling of regular human insulin, insulin aspart, insulin lispro, insulin glulisine, and regular human insulin. This only includes subjects that participated in the Multiplex PK profiling part of the protocol and not the continuous insulin monitoring part of the protocol.
  Multiplex pharmacokinetic profiling
- Continuous Insulin Monitoring Only: Continuous insulin monitoring of insulin lispro. This only includes subjects that participated in the continuous insulin monitoring part of the protocol and did not participate in the Multiplex PK profiling part of the protocol.
  Continuous insulin monitoring
- Both Multiplex PK and Continuous Insulin Monitoring: Participants that enrolled and completed both parts of the trial.
Arm/Group | Multiplex Pharmacokinetic Profiling Only | Continuous Insulin Monitoring Only | Both Multiplex PK and Continuous Insulin Monitoring
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/29 | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes